CLINICAL TRIAL: NCT04961736
Title: Ultrasound Evaluation of Hamstring Tendon Regeneration After Anterior Cruciate Ligament Reconstruction and Its Influence on Gait Touch Information
Brief Title: Ultrasound Evaluation of Hamstring Tendon Regeneration After ACL Reconstruction and Its Influence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OR005
Record Dates: First submitted 2020-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2020-07

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; gait analysis; plantar pressure; Ultrasound evaluation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior Cruciate Ligament injury and reconstruction group: According to the previous clinical diagnosis, volunteers who has never suffered the Anterior Cruciate Ligament injury.
  Interventions: Other: no intervention
- normal control group: According to the previous clinical diagnosis, volunteers who has never suffered the lower extremity sports injuries.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study, with no intervention

SUMMARY:
High incidence rate of knee osteoarthritis and gait analysis are important for early assessment of biomechanics. ACL injury is an ideal clinical model for studying knee osteoarthritis.

To clarify the mechanism between the biomechanical status of knee joint and the change of gait touch information, and to provide scientific basis for quantifying and evaluating the biomechanical status of knee joint in dynamic load-bearing state.

DETAILED DESCRIPTION:
Objective: to analyze the shape and function of the regenerated hamstring tendon within 2 years after the removal of the hamstring tendon in ACL reconstruction, reveal the change rule of the characteristics of hamstring tendon regeneration and its biomechanical changes, and guide the selection of operation and postoperative rehabilitation.

Methods: 55 healthy people and 55 male patients with ACL reconstruction were recruited. All completed the basic rehabilitation training under the guidance of the postoperative rehabilitation program. Using infrared motion capture system, three-dimensional force measuring platform, isokinetic muscle force testing system and ultrasound, the anterior cruciate ligament reconstruction patients were tested before operation, 2 weeks, 3 months, 6 months, 12 months after operation and 24 months after operation.

Outcome evaluation indicators and statistical methods: evaluation indicators: (1) three dimensional motion capture and analysis results: 1) peak ground reaction force; 2) three-dimensional angle and torque of hip, knee and ankle joints in different stages; (2) isokinetic muscle strength results: bilateral knee extension torque and knee flexion torque at different angles and angular velocities. (3)Ultrasound evaluation: the thickness, cross-sectional area and shear wave velocity of the semitendinosus were measured.

Statistical methods: ① repeated measurement analysis of variance (ANOVA) was used to test the effects of different time after operation on the three-dimensional gait characteristics, muscle strength and tendon regeneration characteristics. ② Independent sample t-test was used to test the three-dimensional characteristics, muscle strength and tendon condition of patients at different time points after operation. ③ The difference of three-dimensional gait characteristics, muscle strength and tendon between the healthy side and the affected side at different time points after operation were examined by paired sample t-test. ④ Bivariate correlation analysis was used to analyze whether the thickness, cross-sectional area, shear wave propagation velocity and postoperative time were related.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital.
* With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures).
* All participants have no known disorders or diseases other than ACL rupture.

Exclusion Criteria:

* Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion criteria: Age: 18-35 years old. Patients who have isolated ACL injury and receive ACL reconstruction surgery at Peking University Third Hospital. With isolated ACL injury (an ACL injury with no need for surgical repairs to other knee structures). All participants have no known disorders or diseases other than ACL rupture.
  Exclusion criteria: Female patients who are pregnant, or suspected pregnant, or in breastfeeding will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
peak ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
peak ground reaction force | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
peak ground reaction force | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
peak ground reaction force | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
peak ground reaction force | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of hip in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of hip in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of hip in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of hip in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of hip in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
bilateral knee extension torque | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
bilateral knee extension torque | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
bilateral knee extension torque | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
bilateral knee extension torque | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
bilateral knee extension torque | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
knee flexion torque at different angles | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
knee flexion torque at different angles | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
knee flexion torque at different angles | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
knee flexion torque at different angles | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
knee flexion torque at different angles | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angular velocities | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angular velocities | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angular velocities | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angular velocities | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angular velocities | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
the thickness of the semitendinosus | On the day of enrollment.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | On the day of enrollment.
  Ultrasound evaluation was made by Ultrasonic detector.
the thickness of the semitendinosus | At 2 weeks after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | At 2 weeks after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the thickness of the semitendinosus | At 3 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | At 3 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the thickness of the semitendinosus | At 6 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | At 6 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the thickness of the semitendinosus | At 12 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | At 12 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the thickness of the semitendinosus | At 24 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
the cross-sectional area of the semitendinosus | At 24 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
shear wave velocity of the semitendinosus | On the day of enrollment.
  Ultrasound evaluation was made by Ultrasonic detector.
shear wave velocity of the semitendinosus | At 3 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
shear wave velocity of the semitendinosus | At 6 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
shear wave velocity of the semitendinosus | At 12 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
shear wave velocity of the semitendinosus | At 24 months after Anterior Cruciate Ligament reconstruction.
  Ultrasound evaluation was made by Ultrasonic detector.
torque of hip, knee and ankle joints in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of hip, knee and ankle joints in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of hip, knee and ankle joints in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of hip, knee and ankle joints in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of hip, knee and ankle joints in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of knee joints in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of knee joints in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of knee joints in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of knee joints in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of knee joints in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of ankle joints in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of ankle joints in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of ankle joints in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of ankle joints in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
angle of ankle joints in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of knee joints in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of knee joints in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of knee joints in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of knee joints in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of knee joints in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of ankle joints in different stages | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of ankle joints in different stages | At 3 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of ankle joints in different stages | At 6 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of ankle joints in different stages | At 12 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.
torque of ankle joints in different stages | At 24 months after Anterior Cruciate Ligament reconstruction.
  Three-dimensional gait analysis system and plantar pressure were used during walking, running, cutting and jumping.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | On the day of enrollment, at 3 months, 6 months, 12 months after operation and 24 months after Anterior Cruciate Ligament reconstruction.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No